CLINICAL TRIAL: NCT00410956
Title: A Phase II Study of Hepatic Arterial Infusion With Floxuridine and Dexamethasone in Combination With Intravenous Bevacizumab (A Monoclonal Antibody to Vascular Endothelial Growth Factor-A), in Patients With Unresectable Primary Hepatic Malignancy
Brief Title: Floxuridine and Dexamethasone as a Hepatic Arterial Infusion and Bevacizumab in Treating Patients With Primary Liver Cancer That Cannot be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-114; MSKCC-06114; GENENTECH-MSKCC-06114
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-05

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; adult primary cholangiocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Bevacizumab; Dexamethasone; Floxuridine; Flow Cytometry; Immunoenzyme Techniques; Immunohistochemistry; Immunologic Techniques

ARMS (1):
- UNRESECTABLE PRIMARY HEPATIC MALIGNANCY (Experimental): All patients enrolled in the study will receive HAI FUDR (0.16 mg/kg X pump volume / pump flow rate), Dexamethasone (1 mg/m2/day) and IV Bevacizumab at 5mg/kg. Chemotherapy with HAI FUDR/Dex will commence no sooner than 14 days post surgical placement of HAI pump; patients will receive their first treatment with Bevacizumab no sooner than 28 days post surgical placement of HAI pump.
  Interventions: Biological: bevacizumab; Drug: dexamethasone; Drug: floxuridine; Genetic: protein expression analysis; Other: flow cytometry; Other: immunoenzyme technique; Other: immunohistochemistry staining method; Other: immunologic technique; Other: laboratory biomarker analysis; Procedure: dynamic contrast-enhanced magnetic resonance imaging

INTERVENTIONS:
Biological: bevacizumab
Drug: dexamethasone
Drug: floxuridine
Genetic: protein expression analysis
Other: flow cytometry
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Other: immunologic technique
Other: laboratory biomarker analysis
Procedure: dynamic contrast-enhanced magnetic resonance imaging

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as floxuridine and dexamethasone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving chemotherapy directly into the arteries around the tumor together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving floxuridine and dexamethasone as a hepatic arterial infusion together with bevacizumab works in treating patients with unresectable primary liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the median time to progression in patients with unresectable primary hepatic malignancy treated with hepatic arterial infusion comprising floxuridine and dexamethasone in combination with systemic bevacizumab.

Secondary

* Determine the utility of dynamic contrast-enhanced MRI (DCE-MRI) for assessing changes in tumor perfusion before and during treatment.
* Correlate DCE-MRI findings with radiographic tumor response.

Tertiary

* Correlate the expression patterns of vascular endothelial growth factor (VEGF) receptor (VEGFR)-1, VEGFR-2, and VEGFR-3 and their cognate ligands (including VEGF-A, VEGF-B, VEGF-C, VEGF-D, and placenta growth factor [PlGF]) with disease progression and survival after therapy.
* Assess the pro-angiogenic activity of peripheral blood before and during treatment.
* Assess tumors for immunohistochemical markers of hypoxia (e.g., hypoxia-inducible factor [HIF-1α], carbonic anhydrase IX [CA IX], and glucose transporters [Glut-1 and Glut-3]) for correlation with initial and treatment-related changes in perfusion and permeability, as determined by DCE-MRI.

OUTLINE: This is an open-label, nonrandomized study.

Patients undergo placement of the hepatic arterial infusion (HAI) pump and a cholecystectomy. Approximately 2 weeks later, patients receive floxuridine and dexamethasone by HAI continuously on days 1-14 and bevacizumab IV over 30-90 minutes on day 15 of course 1 and on days 1 and 15 of all subsequent courses. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo dynamic contrast-enhanced MRI (DCE-MRI) on days 1 and 15 of course 1 and then every 8 weeks thereafter.

Tumor and nontumor tissue is collected at the time of the HAI pump placement. Tissue is examined for the expression of vascular endothelial growth factor (VEGF)-A, -B, -C, and -D, placenta growth factor (PlGF), and VEGF receptor (VEGFR)-1, -2, and -3 by immunohistochemistry. Peripheral blood is collected at baseline and on day 1 of each course. Plasma levels of VEGF-A, -B, -C, and -D are measured by immunoenzyme techniques. Blood is also examined by flow cytometry and immunological methods and by protein extraction and analysis of VEGF and VEGFR expression (by western blot). Immunohistochemical markers of hypoxia in tissue, including hypoxia-inducible factor (HIF-1α), carbonic anhydrase IX (CA IX), glucose transporters (Glut-1 and Glut-3), and Ki-67 are assessed.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hepatocellular carcinoma (HCC) or intrahepatic cholangiocarcinoma (ICC)

  * Peripheral, cholangiolar, or cholangiocellular types
  * Mixed HCC/ICC disease allowed
  * Unresectable disease
  * Less than 70% liver involvement
* Radiographically bidimensionally measurable disease, defined as lesion ≥ 2 cm in the greatest diameter
* May have failed prior systemic chemotherapy or ablative therapy
* No radiographic evidence of esophageal varices
* No history of variceal hemorrhage
* No occlusion of the main portal vein or the right and left portal branches
* No clinical ascites
* Patients ineligible for first-line MSKCC protocols for HCC are eligible for this study provided there is no clinical or radiographic evidence of extrahepatic disease
* No metastatic disease, including CNS metastases

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 12 weeks
* Karnofsky performance status 60-100%
* Considered a candidate for general anesthesia and hepatic artery pump placement
* Platelet count > 100,000/mm³
* Albumin > 2.5 g/dL
* Bilirubin < 1.8 mg/dL
* WBC > 3,500/mm³
* PTT < 1.5 times upper limit of normal
* INR < 1.5 OR in-range INR (usually 2.0-3.0) for patients on a stable dose of therapeutic warfarin
* Urine protein < 1+ by dipstick or urine analysis OR urine protein:creatinine ratio < 1.0

  * If proteinuria ≥ 2+ at baseline, patient must have < 1 g protein/24-hour collection
* No concurrent disease or illness that would preclude study participation, including any of the following:

  * Hepatic encephalopathy
  * Sclerosing cholangitis
  * Gilbert's disease
  * Active infection
* No known CNS disease
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab
* No psychiatric illness or social situation that would preclude study compliance
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No serious or nonhealing active wound, ulcer, or bone fracture
* No bleeding diathesis or coagulopathy
* No clinically significant cardiovascular disease, including any of the following:

  * Uncontrolled hypertension, defined as systolic blood pressure (BP) > 150 mm Hg or diastolic BP > 100 mm Hg on antihypertensive medications
  * New York Heart Association class II-IV congestive heart failure
  * Vascular disease (e.g., aortic aneurysm, aortic dissection)
  * Myocardial infarction within the past 6 months
  * Symptomatic peripheral vascular disease
  * Unstable angina within the past 6 months
  * History of hypertensive crisis
  * Transient ischemic attack
  * Stroke
* No other concurrent malignancy except localized basal cell or squamous cell skin cancer
* Chronic hepatitis and/or cirrhosis allowed provided it is Child-Pugh class A disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior and no other concurrent experimental therapy except on a Genentech-sponsored bevacizumab cancer study
* More than 4 weeks since prior major surgical procedure or open biopsy
* More than 1 week since prior minor surgical procedure (e.g., core biopsy), excluding placement of a vascular access device
* No prior external-beam radiation therapy to the liver
* No prior floxuridine
* No chronic daily treatment with nonsteroidal anti-inflammatory medications known to inhibit platelet function
* No chronic daily treatment with aspirin (> 325 mg/day)
* No concurrent or recent use of a thrombolytic agent
* No concurrent major surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-05-09 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William R. Jarnagin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Result] Kemeny NE, Schwartz L, Gonen M, Yopp A, Gultekin D, D'Angelica MI, Fong Y, Haviland D, Gewirtz AN, Allen P, Jarnagin WR. Treating primary liver cancer with hepatic arterial infusion of floxuridine and dexamethasone: does the addition of systemic bevacizumab improve results? Oncology. 2011;80(3-4):153-9. doi: 10.1159/000324704. Epub 2011 Jun 14. PMID 21677464

RESULTS

PARTICIPANT FLOW:
Groups:
- UNRESECTABLE PRIMARY HEPATIC MALIGNANCY: All patients enrolled in the study will receive HAI FUDR (0.16 mg/kg X pump volume / pump flow rate), Dexamethasone (1 mg/m2/day) and IV Bevacizumab at 5mg/kg. Chemotherapy with HAI FUDR/Dex will commence no sooner than 14 days post surgical placement of HAI pump; patients will receive their first treatment with Bevacizumab no sooner than 28 days post surgical placement of HAI pump.
  bevacizumab
  dexamethasone
  floxuridine
  protein expression analysis
  flow cytometry
  immunoenzyme technique
  immunohistochemistry staining method
  immunologic technique
  laboratory biomarker analysis
  dynamic contrast-enhanced magnetic resonance imaging
Period: Overall Study
Arm/Group | UNRESECTABLE PRIMARY HEPATIC MALIGNANCY
Started | 22
Completed | 3
Not Completed | 19
Not completed — Adverse Event | 1
Not completed — Death | 2
Not completed — Lack of Efficacy | 10
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Arm/Group | UNRESECTABLE PRIMARY HEPATIC MALIGNANCY
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 61 [44 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival
Description: Overall median survival from time of initiation of HAI + Bev
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | UNRESECTABLE PRIMARY HEPATIC MALIGNANCY
Number analyzed (Participants) | 22
months | 31.1 [14 to 33.59]

2. Primary Outcome: Median Hepatic Progression Free Survival
Description: Median Hepatic Progression Free Survival. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | UNRESECTABLE PRIMARY HEPATIC MALIGNANCY
Number analyzed (Participants) | 22
months | 11.28 [7.93 to 15.69]

3. Primary Outcome: Median Progression Free Survival
Description: Median Progression Free Survival. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | UNRESECTABLE PRIMARY HEPATIC MALIGNANCY
Number analyzed (Participants) | 22
months | 8.45 [5.53 to 11.05]

4. Primary Outcome: Antitumor Efficacy (Complete and Partial Response, Stable and Progressive Disease)
Description: Antitumor efficacy (complete and partial response, stable and progressive disease). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | UNRESECTABLE PRIMARY HEPATIC MALIGNANCY
Number analyzed (Participants) | 22
Participants
  Partial Response | 7
  Stable Disease | 15

5. Secondary Outcome: Number of Participants Evaluated for Toxicity as Measured by NCI Common Toxicity Criteria
Description: Toxicity as measured by NCI Common Toxicity Criteria
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | UNRESECTABLE PRIMARY HEPATIC MALIGNANCY
Number analyzed (Participants) | 22
Participants | 22

ADVERSE EVENTS:
Time Frame: Up to 36 months
Arm/Group | UNRESECTABLE PRIMARY HEPATIC MALIGNANCY
All-Cause Mortality (participants affected / at risk) | 21/22
Serious Adverse Events (participants affected / at risk) | 12/22
Other Adverse Events (participants affected / at risk) | 17/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UNRESECTABLE PRIMARY HEPATIC MALIGNANCY (N=22)
Pain, headache, nausea (Nervous system disorders) | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1
Chest pain (General disorders) | 1
Mucosal tear, duodenal bulb (Eye disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Portal hypertension, esophageal varices (Hepatobiliary disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
PV thrombosis (Hepatobiliary disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Confusion (Psychiatric disorders) | 1
Myocardial infarct (Cardiac disorders) | 1
Allergic reaction (Immune system disorders) | 1
Ileitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UNRESECTABLE PRIMARY HEPATIC MALIGNANCY (N=22)
Liver function derangement (Hepatobiliary disorders) | 12
Pain (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-12-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT00410956/Prot_SAP_000.pdf